CLINICAL TRIAL: NCT03944954
Title: Neural Mechanisms of Cannabinoid-impaired Decision-Making in Emerging Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michael J. Wesley, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michael J. Wesley, PhD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: K01DA043652 (NIH); K01DA043652 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Neurosciences; Substance-Related Disorders; Behavior Problem
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either excitatory or inhibitory TMS treatment arms. All individuals will receive multiple doses of oral THC (0, 10 and 30mg) and TMS (real or sham).
Who Masked: Investigator
Masking Description: Functionality will be tested following combinations of THC and TMS will be tested in randomized, double-blind, placebo- and sham-controlled experiments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Excitatory TMS (Experimental): Individuals assigned to this group will receive excitatory (real and sham) TMS in combination with 0, 10, and 30mg THC.
  Interventions: Device: Placebo TMS Sham; Drug: Marinol 10Mg Capsule TMS Sham; Drug: Marinol 30Mg Capsule TMS Sham; Device: Placebo TMS Real; Other: Marinol 10Mg Capsule TMS Real; Other: Marinol 30Mg Capsule TMS Real
- Inhibitory TMS (Experimental): Individuals assigned to this group will receive inhibitory (real and sham) TMS in combination with 0, 10, and 30mg THC.
  Interventions: Device: Placebo TMS Sham; Drug: Marinol 10Mg Capsule TMS Sham; Drug: Marinol 30Mg Capsule TMS Sham; Device: Placebo TMS Real; Other: Marinol 10Mg Capsule TMS Real; Other: Marinol 30Mg Capsule TMS Real

INTERVENTIONS:
Device: Placebo TMS Sham — Individuals will receive placebo dose and sham TMS.
  Other Names: Placebo; Sham TMS
Drug: Marinol 10Mg Capsule TMS Sham — Individuals will receive 10mg dose and sham TMS.
  Other Names: 10mg THC; Sham TMS
Drug: Marinol 30Mg Capsule TMS Sham — Individuals will receive 30mg dose and sham TMS.
  Other Names: 30mg THC; Sham TMS
Device: Placebo TMS Real — Individuals will receive placebo and real TMS.
  Other Names: Placebo; Real TMS
Other: Marinol 10Mg Capsule TMS Real — Individuals will receive10mg THC and real TMS. Intervention type: Other (combination device/drug intervention)
  Other Names: 10mg THC; Real TMS
Other: Marinol 30Mg Capsule TMS Real — Individuals will receive 30mg THC and real TMS. Intervention type: Other (combination device/drug intervention)
  Other Names: 30mg THC; Real TMS

SUMMARY:
Emerging adults are a particularly vulnerable group for experiencing the immediate and potentially lifelong negative impacts of habitual cannabis use, and trends suggest that cannabis use disorder (CUD) will soon escalate in this population. The proposed research will combine clinical pharmacology, non-invasive brain stimulation, and neuroimaging techniques to establish the brain mechanisms of cannabinoid-impaired decision-making processes in emerging adults with CUD. Results from this project will inform CUD prevention/treatment efforts in this high-risk group and address a growing public health concern.

DETAILED DESCRIPTION:
This mentored career development award (K01) will enable Dr. Michael J. Wesley to achieve his long-term goal of becoming an independent investigator with a clinical research program examining cannabis use disorder (CUD) in emerging adults, which is a current NIDA funding priority. Dr. Wesley is a new Assistant Professor at the University of Kentucky (UK) College of Medicine. The activities proposed in this award build on Dr. Wesley's background in neuroimaging and drug abuse research and will allow him to accomplish these specific short-term objectives: Become an expert in (1) clinical pharmacology and (2) non-invasive brain stimulation research, and enhance/develop his (3) knowledge of the responsible conduct of research, (4) skills for scientific communication and grant writing, and (5) ability to manage an independent research program. UK has numerous faculty and projects focused on drug abuse research and is an ideal environment for Dr. Wesley to successfully complete this award. Dr. Wesley has assembled a stellar mentoring team consisting of Dr. Josh Lile (Mentor), who runs a successful NIH-funded clinical pharmacology research program at UK and Drs. Mark George (Co-Mentor) and Colleen A. Hanlon of the Brain Stimulation Laboratory at the Medical University of South Carolina, Together they will guide and oversee Dr. Wesley's training in clinical pharmacology, brain stimulation, and scientific communication and grant writing. Dr. Wesley has proposed to engage in a series of formal classes, lab exchanges, and research seminars/meetings that will assist him in accomplishing the objectives of this award.

The proposed research project is novel, innovative, and rigorous. It will combine the acute administration of Δ9-tetrahydrocannabinol (THC), the main psychoactive ingredient in cannabis, with brain stimulation and neuroimaging to examine the role of the dorsal lateral prefrontal cortex (DLPFC) and connected brain areas in drug-impaired decision-making processes. Specifically, transcranial magnetic stimulation (TMS) will be used to raise or lower DLPFC functionality following the administration THC in randomized, double-blind, placebo- and sham-controlled experiments.

Aim 1 will test the hypotheses that excitatory TMS (raising DLPFC functionality) will attenuate the impairing effects of THC on study outcomes.

Aim 2 will test the hypotheses that inhibitory TMS (lowering DLPFC functionality) will enhance the impairing effects of THC on study outcomes.

Results from this project will improve the investigator's understanding of the mechanisms involved in cannabis-impaired decision-making, which will inform CUD management and address a growing public health concern.

ELIGIBILITY:
Inclusion Criteria:

* Habitual cannabis use problems
* Body Mass Index ≤30

Exclusion Criteria:

* Past or current serious physical or mental health
* Sesame seed oil allergy
* Irregular health issues identified by the Study Physician
* Standard magnetic resonance imaging and transcranial magnetic stimulation exclusion criteria (e.g., metal implants, history of epilepsy, etc.)
* Lack of affective form of birth control (females)
* Pregnancy (females)

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Wesley, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Neurobehavioral Systems Lab of the University of Kentucky College of Medicine, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty young adults (N=40; n=20 per Experiment) aged 18-34 who report habitual cannabis use (20 or more days per month) or meet hazardous cannabis use criteria will complete the study. A 15% dropout rate is assumed. Subjects will be matched on sex, age and education. Enrollment will approximate the demographic proportions of Fayette County, KY. so we anticipate enrolling members mostly from those demographic categories.
Groups:
- Excitatory TMS: Combinations of active and placebo THC with real and sham excitatory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real or sham excitatory TMS.
- Inhibitory TMS: Combinations of active and placebo THC with real and sham inhibitory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real and sham inhibitory TMS.
Period: Overall Study
Arm/Group | Excitatory TMS | Inhibitory TMS
Started | 58 | 8
Training Session | 24 | 5
0mg Marinol Sham TMS | 13 | 4
0mg Marinol Real TMS | 14 | 4
10mg Marinol Sham TMS | 13 | 4
10mg Marinol Real TMS | 12 | 4
30mg Marinol Sham TMS | 12 | 5
30mg Marinol Real TMS | 12 | 4
Completed | 11 | 4
Not Completed | 47 | 4
Not completed — Withdrawal by Subject | 22 | 4
Not completed — Lost to Follow-up | 18 | 0
Not completed — Failed Medical Screening | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Excitatory TMS: Combinations of THC and excitatory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real and sham TMS
- Inhibitory TMS: Combinations of THC and inhibitory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real and sham TMS
- Total: Total of all reporting groups
Arm/Group | Excitatory TMS | Inhibitory TMS | Total
Number analyzed (Participants) | 58 | 8 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 8 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (4.5) | 27 (7.0) | 23.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 45 | 5 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 57 | 8 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 1 | 16
  White | 37 | 7 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 58 | 8 | 66

OUTCOME MEASURES:

1. Primary Outcome: Alpha Learning Rate
Description: In a Probabilistic Reinforcement Learning Choice (PRLC) task, two stimuli are presented and choosing either could result in a monetary reinforcer, but the reinforcement probabilities of the stimuli differ, and change throughout the task. Individuals attempt to optimize choices according to learned probabilities and track changing probabilities over time.
  PRLC performance allows mathematical modeling of trial-by-trial data under "real-world" uncertainty and yields computational parameters, such as the learning rate. Choice data were analyzed using a Rescorla-Wanger learning model with an alpha learning rate, beta inverse temperature, and perseveration global parameters. Model-derived learning rates are indicative of an individual's ability to learn from previous choice outcomes to update future decision-making. For this task, learning rates range from 0-1 with lower values indicative of more optimal learning.
Time Frame: Measure collected at 2 time points: Baseline (0HR) and Post TMS Administration (3HR)
Population: Of the 58 total participants assigned to the excitatory TMS condition, 15 individuals completed at least one experimental session.
  Of the 8 total participants assigned to the inhibitory TMS condition, 6 individuals completed at least one experimental session.
Measure: Mean (Standard Deviation); unit: Alpha Coefficient
Arm/Group | Excitatory TMS | Inhibitory TMS
Number analyzed (Participants) | 15 | 6
Alpha Coefficient
  Baseline 0mg Sham: number analyzed (Participants) | 13 | 6
  Baseline 0mg Sham | .62 (.28) | .43 (.37)
  3HR 0mg Sham: number analyzed (Participants) | 13 | 6
  3HR 0mg Sham | .55 (.31) | .21 (.23)
  Baseline 0mg Real: number analyzed (Participants) | 12 | 6
  Baseline 0mg Real | .71 (.27) | .53 (.41)
  3HR 0mg Real: number analyzed (Participants) | 14 | 6
  3HR 0mg Real | .58 (.33) | .48 (.34)
  Baseline 10mg Sham: number analyzed (Participants) | 12 | 6
  Baseline 10mg Sham | .62 (.32) | .49 (.15)
  3HR 10mg Sham: number analyzed (Participants) | 12 | 6
  3HR 10mg Sham | .62 (.28) | .52 (.41)
  Baseline 10mg Real | .63 (.27) | .53 (.38)
  3HR 10mg Real | .63 (.28) | .32 (.38)
  Baseline 30mg Sham | .64 (.29) | .48 (.37)
  3HR 30mg Sham | .60 (.29) | .41 (.30)
  Baseline 30mg Real | .66 (.32) | .24 (.16)
  3HR 30mg Real | .79 (.17) | .30 (.22)

2. Primary Outcome: Self-Report Subjective "High"
Description: A Visual Analogue Scale (VAS) was used to measure the acute subjective effects of THC at varying doses (0mg, 10mg, 30mg). Responses are made for VAS items along a 100-unit scale anchored on the extremes by "Not At All" (0) and "Extremely" (100) with a higher score meaning more of the effect. Participants were instructed to select "Not At All" (0) for all baseline (0HR) measures. Post-TMS administration (real or sham), participant self-reported their subjective "high" on the VAS with higher values indicating a more intense sensation of "high".
Time Frame: Measured 2 times: Baseline (0HR) and 3 hours (3HR) after capsule administration on each drug condition (0mg, 10mg, 30mg)
Population: Of the 58 participants assigned to the Excitatory TMS condition, as max of 14 participants had usable data from at least one experimental session.
  Of the 8 participants assigned to the Inhibitory TMS condition, as max of 4 participants had usable data from at least one experimental session.
Measure: Mean (Standard Deviation); unit: score on a 100pt VAS scale
Groups:
- Excitatory TMS: Combinations of THC and excitatory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive excitatory TMS.
- Inhibitory TMS: Combinations of THC and inhibitory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive inhibitory TMS.
Arm/Group | Excitatory TMS | Inhibitory TMS
Number analyzed (Participants) | 14 | 4
score on a 100pt VAS scale
  "High" 0mg THC Real TMS | 2.9 (5.4) | 0 (0)
  "High" 10mg THC Real TMS: number analyzed (Participants) | 12 | 4
  "High" 10mg THC Real TMS | 13.8 (24.4) | 3.8 (7.5)
  "High" 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  "High" 30mg THC Real TMS | 24.6 (27.3) | 5 (10)
  "High" 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  "High" 0mg THC Sham TMS | 1.2 (2.2) | 3.8 (7.5)
  "High" 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  "High" 10mg THC Sham TMS | 15 (20.3) | 1.3 (2.5)
  "High" 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  "High" 30mg THC Sham TMS | 36.5 (32) | 12.5 (21.8)

3. Primary Outcome: Elasticity of Demand
Description: Elasticity of Demand was measured by the Cannabis Purchase Task (CPT) where participants are asked how many "hits" of cannabis they would consume at 16 different price points in ascending order ($0-$140). Higher elasticity values indicate a greater sensitivity to changing price points resulting in a reduced demand for "hits" of THC at increasing price points.
Time Frame: Measured 2 times: Baseline (0HR) and Post-TMS (3HR) after THC administration on each drug condition (0mg, 10mg, 30mg).
Population: Of the 58 participants assigned to the excitatory TMS condition, 13 individuals had usable data from at least one experimental session.
  Of the 8 participants assigned to the excitatory TMS condition, 4 individuals had usable data from at least one experimental session.
Measure: Mean (Standard Deviation); unit: log(hits per dollar)
Groups:
- Excitatory TMS: Combinations of THC and excitatory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real or sham TMS
- Inhibitory TMS: Combinations of THC and inhibitory TMS.
  Marinol: Individuals will receive 0, 10, 30mg of Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive real or sham TMS
Arm/Group | Excitatory TMS | Inhibitory TMS
Number analyzed (Participants) | 13 | 4
log(hits per dollar)
  Baseline 0mg THC Real TMS: number analyzed (Participants) | 13 | 3
  Baseline 0mg THC Real TMS | .005 (.008) | .004 (.003)
  3HR 0mg THC Real TMS: number analyzed (Participants) | 11 | 4
  3HR 0mg THC Real TMS | .006 (.009) | .007 (.007)
  Baseline 10mg THC Real TMS: number analyzed (Participants) | 10 | 4
  Baseline 10mg THC Real TMS | .005 (.008) | .003 (.002)
  3HR 10mg THC Real TMS: number analyzed (Participants) | 9 | 3
  3HR 10mg THC Real TMS | .006 (.009) | .002 (.001)
  Baseline 30mg THC Real TMS: number analyzed (Participants) | 9 | 2
  Baseline 30mg THC Real TMS | .004 (.002) | .005 (.003)
  3HR 30mg THC Real TMS: number analyzed (Participants) | 9 | 3
  3HR 30mg THC Real TMS | .006 (.008) | .000 (.000)
  Baseline 0mg THC Sham TMS: number analyzed (Participants) | 9 | 4
  Baseline 0mg THC Sham TMS | .005 (.009) | .005 (.006)
  3HR 0mg THC Sham TMS: number analyzed (Participants) | 11 | 4
  3HR 0mg THC Sham TMS | .005 (.009) | .006 (.009)
  Baseline 10mg THC Sham TMS: number analyzed (Participants) | 10 | 3
  Baseline 10mg THC Sham TMS | .006 (.009) | .004 (.002)
  3HR 10mg THC Sham TMS: number analyzed (Participants) | 11 | 4
  3HR 10mg THC Sham TMS | .005 (.009) | .003 (.002)
  Baseline 30mg THC Sham TMS: number analyzed (Participants) | 8 | 2
  Baseline 30mg THC Sham TMS | .004 (.004) | .004 (.004)
  3HR 30mg THC Sham TMS: number analyzed (Participants) | 8 | 4
  3HR 30mg THC Sham TMS | .005 (.006) | .007 (.007)

4. Primary Outcome: Working Memory Performance
Description: Working memory (WM), the ability to hold a finite amount of information for a set amount of time, is measured by the N-Back task. Here, participants were presented with a sequence of letters and must indicate when the letter currently being viewed matches the one from N steps earlier in the sequence. The load factor "N" is adjusted between 0, 1, and 2 to adjust the difficulty of the task (0-Back = no WM load, 1-Back = minimal WM load, 2-Back = greater WM load) where a higher score means better memory performance. Outcomes are reported as the Total Accuracy Percentage (Correct Choices/Total Choices) x 100%
Time Frame: Measured 2 times: Baseline (0HR) and Post-TMS (3HR) after THC administration on each drug condition (0mg, 10mg, 30mg).
Population: Of the 58 participants assigned to the excitatory TMS condition, 14 individuals had usable data from at least one experimental session.
  Of the 8 participants assigned to the excitatory TMS condition, 4 individuals had usable data from at least one experimental session.
Measure: Mean (Standard Deviation); unit: percentage of correct choices
Arm/Group | Excitatory TMS | Inhibitory TMS
Number analyzed (Participants) | 14 | 4
percentage of correct choices
  Baseline 0back 0mg THC Real TMS | 98.0 (1.7) | 96.3 (4.3)
  Baseline 1back 0mg THC Real TMS | 93.0 (4.2) | 90 (12.4)
  Baseline 2back 0mg THC Real TMS | 90.1 (4.7) | 86.3 (21.4)
  Baseline 0back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  Baseline 0back 10mg THC Real TMS | 97.1 (3.4) | 98.3 (1.4)
  Baseline 2back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  Baseline 2back 10mg THC Real TMS | 90.2 (4.9) | 93.3 (7.6)
  Baseline 1back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  Baseline 1back 10mg THC Real TMS | 93.3 (4.3) | 93.3 (3.8)
  Baseline 0back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  Baseline 0back 30mg THC Real TMS | 97.7 (2.2) | 98.1 (1.3)
  Baseline 1back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  Baseline 1back 30mg THC Real TMS | 92.5 (3.68) | 85 (21.7)
  Baseline 2back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  Baseline 2back 30mg THC Real TMS | 89.2 (5.5) | 87.5 (14.3)
  Baseline 0back 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 0back 0mg THC Sham TMS | 98.1 (2.2) | 96.9 (3.2)
  Baseline 1back 0mgTHC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 1back 0mgTHC Sham TMS | 92.1 (4.8) | 89.4 (11.3)
  Baseline 2back 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 2back 0mg THC Sham TMS | 88.3 (4.3) | 85.0 (21.4)
  Baseline 0back 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 0back 10mg THC Sham TMS | 96.4 (3.8) | 93.1 (12.1)
  Baseline 1back 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 1back 10mg THC Sham TMS | 92.1 (4.9) | 92.5 (10.2)
  Baseline 2back 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 2back 10mg THC Sham TMS | 87.9 (6.4) | 83.8 (19.7)
  Baseline 0back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 0back 30mg THC Sham TMS | 96.5 (3.5) | 96.3 (2.5)
  Baseline 1back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 1back 30mg THC Sham TMS | 95 (2.8) | 90.6 (5.5)
  Baseline 2back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  Baseline 2back 30mg THC Sham TMS | 86.9 (6.9) | 87.5 (12.6)
  3HR 0back 0mg THC Real TMS | 97.5 (3.4) | 96.7 (3.2)
  3HR 1back 0mg THC Real TMS | 91.4 (3.1) | 92.5 (3.5)
  3HR 2back 0mg THC Real TMS | 87.3 (5.8) | 89.4 (13.6)
  3HR 0back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  3HR 0back 10mg THC Real TMS | 96.7 (3.1) | 98.3 (1.4)
  3HR 1back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  3HR 1back 10mg THC Real TMS | 92.5 (4.9) | 97.5 (4.3)
  3HR 2back 10mg THC Real TMS: number analyzed (Participants) | 12 | 3
  3HR 2back 10mg THC Real TMS | 87.3 (7.5) | 95 (6.6)
  3HR 0back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  3HR 0back 30mg THC Real TMS | 96.7 (3.6) | 98.1 (2.4)
  3HR 1back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  3HR 1back 30mg THC Real TMS | 88.3 (7.4) | 90.6 (5.2)
  3HR 2back 30mg THC Real TMS: number analyzed (Participants) | 12 | 4
  3HR 2back 30mg THC Real TMS | 86.9 (5.9) | 90.6 (8.8)
  3HR 0back 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 0back 0mg THC Sham TMS | 96.7 (4.1) | 97.5 (2.0)
  3HR 1back 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 1back 0mg THC Sham TMS | 91.7 (5.6) | 93.8 (7.8)
  3HR 2back 0mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 2back 0mg THC Sham TMS | 89.0 (6.0) | 87.5 (10.6)
  3HR 0back 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 0back 10mg THC Sham TMS | 96.2 (3.0) | 90 (18.4)
  3HR 1back 10mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 1back 10mg THC Sham TMS | 92.3 (5.5) | 85.6 (19.1)
  3HR 2back 10mg THC Sham TMS | 88.5 (7.0) | 82.5 (23.8)
  3HR 0back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 0back 30mg THC Sham TMS | 96.7 (3.7) | 94.4 (3.8)
  3HR 1back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 1back 30mg THC Sham TMS | 92.9 (3.2) | 91.3 (7.5)
  3HR 2back 30mg THC Sham TMS: number analyzed (Participants) | 13 | 4
  3HR 2back 30mg THC Sham TMS | 87.3 (8.5) | 87.5 (14.9)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- 0mg Marinol: Marinol: Individuals will receive 0mg Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive either excitatory or inhibitory TMS.
- 10mg Marinol: Marinol: Individuals will receive 10mg Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive either excitatory or inhibitory TMS.
- 30mg Marinol: Marinol: Individuals will receive 30mg Marinol.
  Transcranial Magnetic Stimulation: Individuals will receive either excitatory or inhibitory TMS.
Arm/Group | 0mg Marinol | 10mg Marinol | 30mg Marinol
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 1/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 0/17 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0mg Marinol (N=18) | 10mg Marinol (N=17) | 30mg Marinol (N=17)
Headaches (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — The subject reported headaches attributed to the first experimental administration of TMS. Headaches are noted as potential side effects of TMS in the subject consent form, so this AE was anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03944954/Prot_SAP_ICF_001.pdf